CLINICAL TRIAL: NCT00069485
Title: Evaluation of HIV-Specific Immunological and Virological Responses of HIV-1 Multiply-Exposed Seronegative Individuals
Brief Title: Resistance to HIV Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 5R01AI047086-03 (NIH); 5R01AI047086-03 (NIH)
Record Dates: First submitted 2003-09-26; First posted 2003-09-30 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The immune systems of some individuals may be capable of resisting HIV infection. These individuals do not appear to be infected with HIV despite multiple sexual encounters with HIV infected partners. This study will examine the immune systems of these individuals to determine what factors are responsible for their ability to resist HIV infection.

Study hypothesis: Some long-term, multiply-exposed seronegative persons have relative resistance to HIV infection maintained by T cell responses.

DETAILED DESCRIPTION:
Rare individuals appear naturally resistant to overt HIV-1 infection despite repeated sexual exposures. These individuals, referred to as exposed seronegatives (ES), represent a unique population in which to evaluate mechanisms by which HIV-1 replication is either controlled or aborted. The purpose of the study is to analyze HIV-specific immune responses, both cellular and humoral, that exist in seronegative individuals who have experienced multiple exposures to HIV by sexual contact.

This study will follow participants for 2 years. Participants will have 25 study visits during the study. Assessments will include HIV tests, viral load measurements, CD4 counts, pregnancy tests, and physical exams.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* HIV uninfected
* Repeated exposures to HIV through unprotected sexual intercourse within the 2 years prior to study entry
* Live in the greater Seattle area
* Plan to stay in the greater Seattle area for the 2 years after study entry

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 1995-12

CONTACTS AND LOCATIONS:
Overall Officials: Julie McElrath, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Fred Hutchinson Cancer Research Center / University of Washington HIV Vaccine Trials Unit, Seattle, Washington, United States